CLINICAL TRIAL: NCT04445896
Title: Exploring Patient Responses to Advance Care Planning: A Qualitative Study
Brief Title: The Responses Study
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Princess Alice Hospice (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRAS: 275766
Record Dates: First submitted 2020-03-09; First posted 2020-06-24 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2022-04

CONDITIONS: Advance Care Planning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: Patients with a diagnosis of a life-limiting illness who have previosuly had a discussion with a healthcare professional about the care they would want at the end of life
  Interventions: Other: Qualitative Interview

INTERVENTIONS:
Other: Qualitative Interview — Qualitative Interview to explore thoughts and feelings related to previous discussions around care at end of life

SUMMARY:
The issue Patients who are living with a life-limiting and progressive illness are often encouraged by the healthcare professionals looking after them to undergo a process called Advance Care Planning (ACP). An advance care plan is a written guide of a patient's likes, dislikes, wishes, and the treatments they would want to refuse or the rituals they would want to follow - whether during illness or at the end of life. The planning process helps patients and their relatives think about different scenarios, and the plans that would be used by medical staff if that patient becomes too ill to communicate. ACP discussions can take many forms and are often described as a process.

It is accepted by healthcare professionals that ACP is useful to patients and their relatives. Research has also focussed on the positive nature of ACP, traditionally looking at issues such as how many patients have achieved their wishes and why, what makes ACP possible, and what prevents patients or healthcare professionals from starting these discussions. Some research has also looked at how patients experience the actual process of ACP itself.

However, there has been little research into the effect ACP discussions can have on a patient and their relatives, or how patients react to ACP discussions. As a result, researchers and healthcare professionals do not have a full understanding of the psychological impact on patients and their families, and any resulting changes in patients' outlook, emotional state, family and clinical relationships, and their behaviours.

Learning more about how patients respond to such important and challenging discussions about their care will be vital in improving healthcare professionals' understanding of how best to carry out ACP conversations, and how best to support patients and their relatives following ACP conversations. It is also important to explore not only the benefits of ACP but also the potential downsides or unexpected problems of having such a difficult conversation.

What the investigators will do The aim of this study is to explore how patients are affected by discussions about their future care, and if these discussions affect how patients think or feel in themselves and what they do. The investigators will conduct qualitative interviews with patients living with a life-limiting illness who have already had ACP discussions with a healthcare professional, to explore how and in what ways ACP discussions have affected patients and their families. Qualitative interviews are semi-structured interviews that are designed to explore issues and what these mean to people in-depth, in order to gather rich data that provides insight into a person's perspectives. They are well suited to exploring subjects about which little is yet known, and also subjects which can be sensitive or challenging.

Location of the study, and participation The study will be conducted from Princess Alice Hospice in Surrey, which provides both inpatient and community palliative care services to a large catchment population of approximately 1 million people, in South West London and Surrey.

The investigators aim to recruit 20 participants to represent a broad range of clinical and demographic characteristics, such as age, gender, ethnicity, diagnosis and borough in which they live, in order to explore the experiences of as diverse a group as possible. Participants will be interviewed in a place convenient for them, such as in their home or the Hospice.

Who the investigators are The study will be led by a clinician currently working in Palliative Care, as part of a Masters in Palliative Care, being undertaken at King's College London. The researcher will be supervised at all times by Dr. Katherine Bristowe and Dr. Lisa Brighton, of King's College London, who possess many years of experience in undertaking research among patients living with and dying from advanced disease, and their families.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and over
2. A palliative care diagnosis confirmed by a referring healthcare professional, i.e. a diagnosis of a life-threatening or life-limiting illness
3. Have completed one or multiple ACP discussions as defined below, at any time prior to referral to study, with a healthcare professional
4. Sufficient cognitive capacity to provide informed consent and complete an interview

For the purposes of recruitment for this study, ACP is defined as:

Any significant discussion with a healthcare professional where patients have discussed their values, goals or preferences for future care. These can include discussions about wishes for further disease-modifying treatment, wishes for intensity of general medical care, preferred places of care and death, discussions around resuscitation and transfer to hospital, and completion of advanced directives. Healthcare professionals can include any doctor, nurse or allied health professional.

Exclusion Criteria:

1. Any patient the researcher has ever met or cared for in a clinical capacity, or knows in any other capacity
2. Any patient who has only had ACP discussions with a volunteer (trained or untrained) or non-healthcare professional
3. Inability to provide informed consent
4. Any patient deemed by the referring healthcare professional to be potentially too unwell or frail to undertake an interview

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from Princess Alice Hospice. Princess Alice is a large Hospice in Surrey which provides inpatient, day services and community services to 9 boroughs in South London, Surrey and Middlesex, with a catchment population of approximately 1 million people. Community home visit and outpatient services are provided by a Consultant led, multi-disciplinary team, and provide care to approximately 850 patients at any one time. Princess Alice has a 20 bedded Palliative Medicine inpatient unit and accepts referrals for symptom control and terminal care admissions, with a typical length of stay of 7-10 days.
  Patients are referred to Princess Alice Hospice for Specialist Palliative Care if they have a diagnosis of a life-limiting or life-threatening disease. Princess Alice Hospice provides holistic palliative care that is aimed to provide physical, psychological, spiritual and social support.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Themes emerging from Qualitative Interview | Throughout study completion, estimated to be 1 year
  Key themes and concepts that emerge from multiple participants qualitative interviews that describe their experiences

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bristowe, PhD, Principal Investigator — King's College London
Locations (1):
- Princess Alice Hospice, Esher, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No